CLINICAL TRIAL: NCT01547858
Title: A Cross-Sectional Study of Hematotoxicity in Workers Exposed to Formaldehyde
Brief Title: Studying Blood Toxicity in Workers Exposed to Formaldehyde
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912055; 12-C-N055
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Blood; Chemical Industry
Keywords: Hematotoxicity; Formaldehyde; Cross-Sectional Study; Occupational Exposure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, buffy coat/Red blood cell, whole blood in PAXgene, Urine, Buccal rinse, Buccal scrape.

SUMMARY:
Background:

- Formaldehyde has many uses in industry and medicine. However, exposure to formaldehyde has been associated with increased risk for myeloid leukemia. There are still questions about how the chemical reacts with bone marrow to increase this cancer risk. Some smaller studies have looked at how it affects stem cells, which are found in bone marrow. Researchers want to develop a much larger study of workers in China. The study will look at different levels of formaldehyde exposure. It will focus on how the chemical affects the blood cells and bone marrow.

Objectives:

- To study the effects of formaldehyde exposure on blood cells and bone marrow.

Eligibility:

- Individuals between 18 and 60 years of age who work in selected factories in Guangdong Province, China.

Design:

* Participants will be screened with a physical exam and medical history. They will also be screened with a work history. Those who have been exposed to benzene, butadiene, styrene, or radiation will not be included.
* Participants will be studied based on their regular formaldehyde exposure level. One-third will be those exposed to more than 1 part per million (ppm) of the chemical. One-third will be those exposed to 0.3 to 1 ppm. A control group will have no exposure to formaldehyde or any other known toxic chemical.
* Participants will provide blood and cheek swab samples. They will also answer questions about their work habits.
* To look at chemical exposure levels, participants will wear a small monitor to work on 3 different days. They may provide additional blood and cell samples as directed.
* No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
Research in industrial workers and professionals exposed to formaldehyde suggests that occupational exposure to this important chemical is associated with increased risk for myeloid leukemia. However, there is still uncertainty about the biologic plausibility of the association because of questions regarding the ability of formaldehyde, which is extremely reactive, to directly or indirectly cause toxicity to the bone marrow. There have been several relatively small studies of the impact of occupational formaldehyde exposure on peripheral blood cells that found some evidence that peripheral blood cells of the myeloid lineage (i.e., granulocytes, platelets) were significantly decreased in exposed workers. We propose to follow-up these findings in a relatively large study population in China. We will study hematologic parameters in 240 higher exposed workers (>1 ppm), 240 workers exposed to lower levels of formaldehyde (0.3 to 1 ppm), and a group of 240 unexposed controls frequency-matched to exposed workers. This study will make an important contribution to our understanding of the leukemogenic potential of formaldehyde, which has important public health and regulatory implications.

ELIGIBILITY:
* INCLUSION CRITERIA:
* The eligible age range for the study will be 18 to 60 years old

EXCLUSION CRITERIA:

Exclusion criteria for both formaldehyde-exposed and control workers will be:

- A history of cancer, chemotherapy, and/or radiotherapy, as well as previous or current occupational exposure to benzene, butadiene, styrene and radiation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will identify formaldehyde-exposed manufacturing workers during the cross-sectional study. The exposed workers have to have held the same job for at least 3 months in the same factory. We expect that the age and sex distribution will be similar in the lower and higher exposed workers. We will enroll controls without previous occupational exposure to formaldehyde or any other genotoxic, hematotoxic or immunotoxic chemicals in two factories that manufacture clothes located in the same@@@geographic area as the utensil producing factories.
Sampling Method: Non-Probability Sample
Enrollment: 708 (Actual)
Dates: Start 2012-02-09 (Actual); Primary Completion 2013-05-30 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Hematotoxicity Change | 2012-2024
  Complete blood counts
Immune Function | 2012- 2024
  immune biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Qing Lan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Guangdong National Poison Control Center (NPCC), Guangzhour, China

REFERENCES:
- [Background] Coggon D, Harris EC, Poole J, Palmer KT. Extended follow-up of a cohort of british chemical workers exposed to formaldehyde. J Natl Cancer Inst. 2003 Nov 5;95(21):1608-15. doi: 10.1093/jnci/djg046. PMID 14600093
- [Background] Hauptmann M, Stewart PA, Lubin JH, Beane Freeman LE, Hornung RW, Herrick RF, Hoover RN, Fraumeni JF Jr, Blair A, Hayes RB. Mortality from lymphohematopoietic malignancies and brain cancer among embalmers exposed to formaldehyde. J Natl Cancer Inst. 2009 Dec 16;101(24):1696-708. doi: 10.1093/jnci/djp416. PMID 19933446
- [Background] Pinkerton LE, Hein MJ, Stayner LT. Mortality among a cohort of garment workers exposed to formaldehyde: an update. Occup Environ Med. 2004 Mar;61(3):193-200. doi: 10.1136/oem.2003.007476. PMID 14985513